CLINICAL TRIAL: NCT01336985
Title: Phase Ib Study of the Safety and Pharmacokinetics of Chemoembolization With Irinotecan-Eluting Beads for the Treatment of Hepatic Metastases
Brief Title: Safety and Pharmacokinetics of Treating Liver Cancer With Drug-Eluting Beads
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 110131; 11-CC-0131
Record Dates: First submitted 2011-04-14; First posted 2011-04-18 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2014-11-03

CONDITIONS: Neoplasm Metastases; Melanoma; Colorectal Neoplasms
Keywords: Chemoembolization; Hepatic Metastases; Irinotecan; Drug Eluding Beads; Colorectal Cancer; Liver Cancer; Hepatic Cancer; Melanoma
MeSH Terms: conditions — Neoplasm Metastasis; Melanoma; Colorectal Neoplasms; Liver Neoplasms | interventions — Irinotecan; Chemoembolization, Therapeutic; Biopsy

INTERVENTIONS:
Drug: Irinotecan
Procedure: Chemoembolization
Device: Drug-Eluting Beads
Procedure: Biopsy

SUMMARY:
Background:

* Cancers in other parts of the body often spread to the liver, developing tumors which in many instances cannot be removed with surgery. Liver chemoembolization is a treatment that is routinely performed to control liver tumors in those who cannot have surgery. It has been shown to prolong survival, but does not cure the cancer. During chemoembolization very tiny beads (drug-eluting beads, or DEB) containing chemotherapy drugs (usually doxorubicin) are administered directly into the blood vessels of a liver tumor. The drug within the beads is then released into the tumor whilethe beads temporarily interrupt the tumor s blood supply.
* Irinotecan, a drug commonly given intravenously to treat colon cancer, has been given in chemoembolization procedures in four other studies that have shown that the treatment is generally well tolerated. Researchers are interested in determining whether giving the drug irinotecan directly into the liver using drug-eluting beads is not only well tolerated but also provides a larger dose directly to the tumor as determined by tumor and normal liver tissue biopsies. The liver biopsies are an optional portion of the study.

Objectives:

- To evaluate the safety and effectiveness of chemoembolization with irinotecan for tumors caused by cancer that has spread to the liver.

Eligibility:

- Individuals at least 18 years of age who have melanoma, colon, or another intra-abdominal cancer that has spread to the liver.

Design:

* Participants will be screened with a physical examination, medical history, blood tests, tumor imaging studies, and liver biopsies.
* Participants will receive up to 3 DEB chemoembolization treatments about 6 weeks apart.
* After two treatments, participants will have imaging studies to see if the tumors have shrunk, and those whose tumors have shrunk may have a third treatment.
* Multiple liver biopsies may be performed and blood samples will be taken to determine how much drug is in the tumor and the circulation, and to see how the tumor reacts to the drug.
* Participants will return for followup visits for up to 1 year....

DETAILED DESCRIPTION:
Background:

* Clinical evidence suggests that hepatic chemoembolization may prolong survival in patients with hepatic metastases.
* Early studies have indicated that chemoembolization using irinotecan drug eluting beads may be more effective in treating hepatic metastases from colon or melanoma primary tumors.

Objectives:

* Primary Objective:

  --To determine the safety of hepatic chemoembolization with drug-eluting beads containing 100mg of irinotecan
* Secondary Objectives:

  * To determine the serum pharmacokinetics and tumor tissue concentrations achieved following hepatic chemoembolization with irinotecan-eluting beads

Eligibility:

* Patients > 18 years of age with pathologically proven hepatic metastases from the gastrointestinal tract, or melanoma with unresectable hepatic lesions.
* Patients whose extent of hepatic metastases represents <60% of total liver volume AND whose extrahepatic metastatic disease is determined to be minimal
* Patients must be ECOG performance status of less than or equal to 2 and a life expectancy of more than 3 months.
* Patients must have adequate organ function.
* Patients must not have had chemotherapy, radiation therapy, or biological therapy for at least 4 weeks prior to starting study treatments.
* Patients are not to receive conventional chemotherapy or therapeutic monoclonal antibodies while on study.
* Patients must not have an acute, critical illness.

Design:

* A Phase Ib trial in which patients undergo hepatic chemoembolization with drug-eluting beads containing 100mg irinotecan.
* Up to 15 patients will be enrolled over 1 year to accrue 10 evaluable patients.
* Patients will undergo up to 3 chemoembolizations.
* Following chemoembolization, patients will have serial serum pharmacokinetic samples drawn and tumor biopsies in order to measure serum and tumor tissue concentrations of irinotecan
* Patients will be followed for one year after completion of the last treatment.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Patients with pathologically proven hepatic-dominant metastases from abdominal or gastrointestinal tract primary malignancy or melanoma where the life limiting component of the disease is hepatic metastasis
* Patients must have unresectable hepatic lesions or must be unable or unwilling to undergo surgical resection. Patients may have undergone prior wedge resection of the liver for metastatic disease
* All patients must be refractory to or intolerant of approved standard systemic therapy.

Specifically:

* Patients with metastatic colorectal must have received 5-FU and leucovorin in combination with either oxaliplatin and/or irinotecan, since level 1 evidence support increase survival with these regimens, compared to 5-FU and leucovorin alone.
* Patients with melanoma must have received IL-2 or other immunotherapy options (such as ipilimumab or adoptive cell therapy) that have been reported to have efficacy.

  * Patients with extrahepatic metastases or an unresected primary lesion will be considered eligible if the extrahepatic disease is minimal
  * Extent of hepatic metastases is <60% of total hepatic volume.
  * Patients must have at least one lesion that can be readily biopsied (at least 10mm diameter)
  * ECOG performance status less than or equal to 2
  * Life expectancy > 3 months
  * At least 18 years of age
  * Age < 85 years
  * Patients must have had no chemotherapy, radiotherapy, or biologic therapy for their malignancy for at least 4 weeks (or until response can be adequately assessed) prior to treatment and must have recovered from all clinically significant side effects of therapeutic and diagnostic interventions. Anti-VEGF agents (eg, Avastin) may not be administered less than 4 weeks prior to DEB-TACE treatment.
  * Patients are not to receive conventional chemotherapy or therapeutic monoclonal antibodies while receiving protocol treatment
  * Hematology:
* Absolute neutrophil count greater than 1500/mm(3) without the support of Filgrastim.
* Platelet count greater than 75,000/mm(3).
* Hemoglobin greater than 8.0 g/dl.

  -Chemistry:
* Serum ALT/AST less than or equal to 3 times the upper limit of normal.
* Serum creatinine less than or equal to 2.0 mg/dl unless the measured creatinine clearance is greater than 60 mL/min
* Total bilirubin less than or equal to 2 mg/dl.
* INR <1.5
* PTT less than or equal to 1.3 times control unless a mixing study confirms the presence of a lupus anticoagulant as the cause for the prolonged PTT.

  * Screening electrocardiogram is normal with QTc less than or equal to 480msec).

EXCLUSION CRITERIA:

* Significant cardiac or pulmonary insufficiency as evidenced by

  * history of congestive heart failure with an LVEF < 40%
  * history of COPD or other chronic pulmonary disease with PFT s indicating an FEV1 less than 30% or a DLCO less than 40% predicted for age
* Portal Vein Occlusion or other contraindications to chemoembolization
* Inflammatory bowel disease
* Prior chemoembolization therapy
* Prior precutaneous hepatic perfusion therapy
* Prior selective internal radiation therapy (SIRT) with Yttrium-90
* Prior biliary diversion surgery
* Previous liver resection other than wedge resection.
* Pregnant patients and nursing mothers will be excluded because of the unknown effects of this therapy on the fetus or nursing infants.
* Patients taking immunosuppressive drugs or requiring ongoing chronic anticoagulation will not be eligible.
* Patients with active bacterial infections with systemic manifestations (malaise, fever, leucocytosis) are not eligible until completion of appropriate therapy.
* Patients with severe allergic reactions to iodine contrast which cannot be controlled by premedication with antihistamines and steroids are not eligible as a hepatic angiogram is needed for this procedure.
* Patients with a known prior hypersensitivity reaction or other contraindication to irinotecan will be excluded.
* Patients taking phenytoin, phenobarbital, carbamazepine, rifampin, rifabutin, St. John s Wort, or other CYP3A inducers or inhibitors are not eligible for this study.
* Patients are prohibited from receiving other experimental agents/adjuvant treatments during the study.
* Patients with more than one active primary malignancy, except for basal cell carcinoma or superficial bladder neoplasia, are to be excluded.

Ages: 18 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2011-03-28; Study Completion 2011-03-28 (Actual)

PRIMARY OUTCOMES:
To determine the safety of hepatic chemoembolization with drug-eluting beads containing 100mg of irinotecan

SECONDARY OUTCOMES:
To determine the serum pharmacokinetics and tumor tissue concentrations achieved following hepatic chemoembolization with irinotecan-eluting beads

CONTACTS AND LOCATIONS:
Overall Officials: Elliot B Levy, M.D., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Adam R, Delvart V, Pascal G, Valeanu A, Castaing D, Azoulay D, Giacchetti S, Paule B, Kunstlinger F, Ghemard O, Levi F, Bismuth H. Rescue surgery for unresectable colorectal liver metastases downstaged by chemotherapy: a model to predict long-term survival. Ann Surg. 2004 Oct;240(4):644-57; discussion 657-8. doi: 10.1097/01.sla.0000141198.92114.f6. PMID 15383792
- [Background] Adam R. Chemotherapy and surgery: new perspectives on the treatment of unresectable liver metastases. Ann Oncol. 2003;14 Suppl 2:ii13-6. doi: 10.1093/annonc/mdg731. PMID 12810452
- [Background] Aliberti C, Tilli M, Benea G, Fiorentini G. Trans-arterial chemoembolization (TACE) of liver metastases from colorectal cancer using irinotecan-eluting beads: preliminary results. Anticancer Res. 2006 Sep-Oct;26(5B):3793-5. PMID 17094403